CLINICAL TRIAL: NCT00383175
Title: Reading Fluency and Accommodative Lag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: R. Kleinstein and J. Sims, UAB
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: F060328003; EY008893 (Other Grant/Funding Number: NEI)
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Ocular Accommodation
Keywords: Ocular Accommodation; Reading

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Autorefractor, standard clinical instrument — Autorefractor, standard clinical instrument was used to assess the children's focusing power at near.

SUMMARY:
The purpose of this study is to determine whether special reading glasses improve children's ability to learn to read.

DETAILED DESCRIPTION:
Many children are believed to under accommodate (have a lag of accommodation) when looking at near targets. If this occurs, the retinal image is out of focus. Children who have a lag of accommodation may have difficulty in focusing their eyes at near for long periods of time. This difficulty could reduce their ability to read fluently. Children with above average lags of accommodation will be randomly assigned to a group which receives special reading glasses or a group which does not. The groups will be assessed using a standard test for reading fluency.

ELIGIBILITY:
Inclusion Criteria:

* Children in grades 1, 2 and 3 who consent and assent to participate

Exclusion Criteria:

* Children in the special education program
* Children who are unwilling to have their eyes dilated or be tested
* Children who are unwilling to wear the glasses

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
DIBELS test scores . | 1 -2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kleinstein, OD,MPH,PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Eutaw Primary School, Eutaw, Alabama, United States